CLINICAL TRIAL: NCT03453515
Title: Reducing HIV Risk Among Adolescents: Evaluating HEART for Teens
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: North Carolina State University (Other)
Responsible Party: Principal Investigator, Laura Widman, Assistant Professor, North Carolina State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: NCState
Record Dates: First submitted 2018-02-27; First posted 2018-03-05 (Actual); Results first posted 2020-09-29 (Actual); Last update posted 2020-09-29 (Actual); Status verified 2020-09

CONDITIONS: HIV Infections; Sexually Transmitted Diseases
MeSH Terms: conditions — HIV Infections; Sexually Transmitted Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HEART (Experimental): Interactive website with five modules to address safer sex motivation, knowledge, attitudes/norms, self-efficacy, and sexual communication skills. Program takes approximately 30-45 minutes to complete.
  Interventions: Behavioral: HEART
- Growing Minds (Other): Attention-matched control website with five modules to address an introduction to mindsets, growth mindsets of intelligence, growth mindsets of self-control, growth mindsets of people, and an integrative summary. Program takes approximately 30-45 minutes to complete.
  Interventions: Behavioral: Growing Minds

INTERVENTIONS:
Behavioral: HEART — Interactive web-based intervention with five modules: motivation, knowledge, attitudes/norms, self-efficacy, and sexual communication skills.
  Arms: HEART
Behavioral: Growing Minds — Interactive web-based intervention with five modules: mindsets introduction, growth mindsets of intelligence, growth mindsets of self-control, growth mindsets of people, and integrative summary.
  Arms: Growing Minds

SUMMARY:
This study evaluates an educational web-based intervention designed to increase adolescent boys' and girls' motivation and skills to engage in safer sexual behavior (HEART: Health Education and Relationship Training). Half of participants will receive HEART and half of participants will receive Growing Minds, an attention-matched control website focused on growth mindsets of intelligence and self-regulation. The ultimate goal of this work is to help youth reduce their risk of HIV and other sexually transmitted diseases and to avoid unplanned pregnancies.

DETAILED DESCRIPTION:
This study evaluates an educational web-based intervention designed to increase adolescent boys' and girls' motivation and skills to engage in safer sexual behavior (HEART: Health Education and Relationship Training). Half of participants will receive HEART and half of participants will receive Growing Minds, an attention-matched control website focused on growth mindsets of intelligence and self-regulation. The ultimate goal of this work is to help youth reduce their risk of HIV and other sexually transmitted diseases and to avoid unplanned pregnancies.

Primary outcomes for this study include 1) acceptability of the program, 2) safer sex self-efficacy, and 3) safer sex intentions.

ELIGIBILITY:
Inclusion Criteria:

* 10th or 11th grader
* Able to read English

Exclusion Criteria:

* None

Ages: 14 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 226 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2018-04-30 (Actual); Study Completion 2019-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Laura Widman, PhD, Principal Investigator — North Carolina State University
Locations (1):
- North Carolina State University, Raleigh, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | HEART | Growing Minds
Started | 113 | 113
Completed | 107 | 100
Not Completed | 6 | 13

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | HEART | Growing Minds | Total
Number analyzed (Participants) | 113 | 113 | 226
Age, Continuous [Mean (Standard Deviation); unit: Years] | 16.27 (.79) | 16.24 (.74) | 16.25 (.76)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 69 | 67 | 136
  Male | 44 | 46 | 90
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 46 | 57 | 103
  Black | 32 | 23 | 55
  Latinx | 28 | 29 | 57
  Other | 7 | 4 | 11
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 113 | 113 | 226
Free/reduced price lunch [Count of Participants; unit: Participants] | 59 | 53 | 112

OUTCOME MEASURES:

1. Primary Outcome: Acceptability
Description: 6-item self-report of program acceptability. Each item analyzed separately for the percentage endorsement. Items were as follows: Liked the program Learned new things Program kept attention Will use information in the future Useful for girls my age Useful for boys my age
  Below we report results for the first item: number of participants who agree that they like the program
Time Frame: immediate post-test at completion of intervention
Population: 7 participants from HEART and 15 participants from Growing Minds did not complete the acceptability questionnaire.
Measure: Count of Participants; unit: Participants
Arm/Group | HEART | Growing Minds
Number analyzed (Participants) | 106 | 98
Participants | 88 | 83

2. Secondary Outcome: HIV/STD Knowledge
Description: HIV/STD knowledge was assessed with 9 items (e.g., "STDs usually have noticeable symptoms, like itching or burning"). These were adapted from previous sexual health knowledge questionnaires (Brown, DiClemente, & Park, 1992; Morton, Nelson, Walsh, Zimmerman, & Coe, 1996) and were used in our previous work (Widman, Golin, et al., 2018). Participants rated each item as True, False, or Don't Know. Responses were recoded as 0 (Incorrect or Don't Know) or 1 (Correct). Scores were summed to reflect the total number of correct HIV/STD knowledge questions (possible range=0-9).
Time Frame: immediate post-test at completion of intervention
Population: 6 participants from HEART and 13 participants from Growing Minds did not complete the HIV/STD knowledge scale at post-test
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | HEART | Growing Minds
Number analyzed (Participants) | 107 | 100
units on a scale | 7.68 (1.79) | 5.74 (1.86)

3. Secondary Outcome: Condom Beliefs
Description: Participants' attitudes about condoms were assessed with the 3-item Effect on Sexual Experiences subscale of the Condom Attitudes Scale Adolescent Version (St. Lawrence et al., 1994). An example item includes, "Condoms take away the pleasure of sex." Responses were on a scale from 1 (Strongly Disagree) to 5 (Strongly Agree; alpha=.77). A mean of the three items was computed, such that higher scores indicate better outcomes (possible range 1-5).
Time Frame: immediate post-test at completion of intervention
Population: 6 participants from HEART and 13 participants from Growing Minds did not complete the condom beliefs scale at post-test
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | HEART | Growing Minds
Number analyzed (Participants) | 107 | 100
units on a scale | 3.85 (.96) | 3.22 (.94)

4. Secondary Outcome: Sexual Assertiveness
Description: Self-reported sexual assertiveness was assessed with 3-items from the Multidimensional Sexual Self-Concept Scale (Snell, 1998). Items such as, "I'm very assertive about the sexual aspects of my life," were rated on a scale from 1 (Strongly Disagree) to 5 (Strongly Agree; alpha=.75). A mean of the three items was computed, such that higher scores indicate better outcomes (possible range 1-5).
Time Frame: immediate post-test at completion of intervention
Population: 6 participants from HEART and 13 participants from Growing Minds did not complete the sexual assertiveness scale at post-test
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | HEART | Growing Minds
Number analyzed (Participants) | 107 | 100
units on a scale | 3.88 (.98) | 3.68 (.75)

5. Secondary Outcome: Safer Sex Intentions
Description: Intentions to discuss sexual health was assessed with a item developed by our research team based on items from the AIDS Risk Behavior Survey (Donenberg, Emerson, Bryant, Wilson, & Weber-Shifrin, 2001) and our previous work (Widman, Golin, et al., 2018). This item asked how likely teens were to discuss sexual health issues, including pregnancy and STDs, with their partner(s) prior to sexual activity (communication intentions). Response options ranged from 1 (not at all likely) to 5 (very likely). Higher scores indicate better outcomes.
Time Frame: immediate post-test at completion of intervention
Population: 6 participants from HEART and 13 participants from Growing Minds did not complete the safer sex intentions item at post-test
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | HEART | Growing Minds
Number analyzed (Participants) | 107 | 100
units on a scale | 4.43 (.83) | 3.97 (1.15)

6. Secondary Outcome: Safer Sex Self-Efficacy
Description: The Self-Efficacy for HIV Prevention Scale (Brown et al., 2014) was used to assess self-efficacy about communication and condom use. Six items assessed confidence communicating about sexual topics (e.g., "How sure are you that you could talk to your partner about safer sex?"). Two items assessed confidence obtaining and using condoms (e.g., "How sure are you that you could have condoms available when you need them?"). Participants responded from 1 (Couldn't do it) to 4 (Very Sure). A mean of all items was computed, such that higher scores indicate better outcomes (possible range 1-4; alpha=.79).
Time Frame: immediate post-test at completion of intervention
Population: 6 participants from HEART and 13 participants from Growing Minds did not complete the safer sex self-efficacy scale item at post-test
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | HEART | Growing Minds
Number analyzed (Participants) | 107 | 100
units on a scale | 3.30 (.66) | 3.21 (.56)

ADVERSE EVENTS:
Time Frame: 1 yr
Arm/Group | HEART | Growing Minds
All-Cause Mortality (participants affected / at risk) | 0/113 | 0/113
Serious Adverse Events (participants affected / at risk) | 0/113 | 0/113
Other Adverse Events (participants affected / at risk) | 0/113 | 0/113

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-10-16): https://cdn.clinicaltrials.gov/large-docs/15/NCT03453515/Prot_SAP_000.pdf